CLINICAL TRIAL: NCT05124431
Title: Single Arm, Single Center, Prospective, Phase II Clinical Study of Anlotinib Hydrochloride Capsule Combined With Everolimus in the First-line Treatment of Advanced Non Clear Cell Renal Cell Carcinoma
Brief Title: Anlotinib Plus Everolimus as First-line Treatment for Advanced Non Clear Cell Renal Cell Carcinoma
Acronym: ALTER-UC-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-37-2340
Record Dates: First submitted 2021-10-15; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma,RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride+Everolimus (Experimental): Anlotinib hydrochloride: ,12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Everolimus:5mg po. qd in 21-day cycle
  Interventions: Drug: Anlotinib hydrochloride; Drug: everolimus

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor.
Drug: everolimus — 5mg po，qd

SUMMARY:
This is a single-centre, single-arm, phase 2 study to evaluate the efficacy and safety of anlotinib hydrochloride plus everolimus in patients with advanced non clear renal cell carcinoma as first-line treatment.

DETAILED DESCRIPTION:
This is a single-arm, phase II trial in non-clear renal cell carcinoma patients. The purpose of this trial is to evaluate the safety and efficacy of anlotinib hydrochloride combined with everolimus in patients with no systematic treatment advanced non clear renal cell carcinoma.

The primary objective: Overall Response Rate(ORR)(according to RECIST version 1.1). The second objectives: progression free survival (PFS), disease control rate (DCR), Overall Survival(OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent, with good compliance
2. Over 18 years
3. ECOG PS:0-1,Life expectancy of more than 6 months
4. Patients with histologically confirmed advanced non-clear renal cell carcinoma. advanced disease is defined as IV(TNM), not available for surgery, locally recurrent or metastatic renal cell carcinoma
5. Did not receive systematic drug treatment for advanced disease.
6. With measurable disease (using RECIST1.1)
7. Main organs function is normal
8. Patients of child-bearing period agree to use appropriate contraception. The serum pregnancy test of women in childbearing period was negative within 4 weeks before enrollment

Exclusion Criteria:

1. History of allergy or intolerance to study drug components;
2. Previously received strong CYP3A4 inhibitor treatment within one week before enrollment or strong CYP3A4 inducer treatment within two weeks before participating in the study.
3. Combined disease / medical history

   1. Clinically significant hemoptysis (more than 50ml of hemoptysis per day) occurred within 3 months before enrollment; or significant clinically significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood at baseline and above , Or suffer from vasculitis, etc.;
   2. Arteriovenous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to pre-chemotherapy, except those who have been cured by the investigator ) And pulmonary embolism, etc.;
   3. Hypertension, and can not be well controlled by antihypertensive drugs (systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg); within 6 months before enrollment, the following conditions occurred: myocardial infarction, severe/unstable angina, NYHA Grade 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure;
   4. Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (such as diabetes, pulmonary fibrosis, acute pneumonia, etc.);
   5. Renal insufficiency: Urine routine test indicates urine protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
   6. The history of live attenuated vaccine vaccination within 28 days before the first study medication or the expected live attenuated vaccine vaccination during the study period;
   7. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis (hepatitis B, defined as HBV-DNA ≥500 IU/ml; hepatitis C, defined as HCV-RNA Higher than the detection limit of the analytical method) or combined with hepatitis B and C co-infection;
   8. Severe infections 4 weeks before the first administration including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc. Active infections with CTCAE ≥ grade 2 requiring systemic antibiotic treatment within 2 weeks before the first administration, Or, during the screening period/before the first administration, fever of unknown origin> 38.5°C (according to the judgment of the investigator, fever caused by tumor can be included in the group); there is evidence of active tuberculosis infection within 1 year before the administration;
   9. Any other malignant tumor was diagnosed within 3 years before entering the study, except for fully treated basal cell carcinoma or squamous cell skin cancer or cervical carcinoma in situ;
   10. Major surgery was performed within 28 days before enrollment (tissue biopsy required for diagnosis and central venous catheter insertion via peripheral venous puncture [PICC] are allowed);
   11. Patients who have had previous organ transplants (except autologous hematopoietic stem cell transplants);
   12. Peripheral neuropathy ≥ Grade 2; patients with active brain metastasis, cancerous meningitis, spinal cord compression, or those with brain or pia mater detected on imaging CT or MRI at the time of screening (treatment has been completed 14 days before enrollment with symptoms Patients with stable brain metastases can be included in the group, but they need to be evaluated by MRI, CT or venography to confirm that they have no symptoms of cerebral hemorrhage);
   13. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction with significant clinical significance.
4. Pregnant or lactating women.
5. Had other serious physical or mental diseases or abnormal laboratory finding,may increase the risk of the study or interfere with the results of the study
6. Patients are unsuitable for the enrollment according to investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to approximately 24 months
  ORR was defined as the percentage of participants in the analysis population who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on investigator evaluation.

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to approximately 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD)
Progression free survival (PFS) | up to approximately 24 months
  The PFS time is defined as time from randomization to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of: "death", "last tumor assessment", "last follow up date" or "last date in drug log"
Overall Survival (OS) | up to approximately 24 months
  OS was defined as time from date of randomization to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Hailiang Zhang, M.D, Study Chair — Fudan University
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China